CLINICAL TRIAL: NCT04276948
Title: Effects of NAD3 Supplementation on Biomarkers of Anti-Aging in Healthy Men and Women
Brief Title: Effects of NAD3 Supplementation on Biomarkers of Aging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Center for Applied Health Sciences, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CS-01-2020
Record Dates: First submitted 2020-02-17; First posted 2020-02-19 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2020-02

CONDITIONS: Aging
Keywords: dietary supplement

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active1 (Experimental): 312 mg dose of active
  Interventions: Dietary Supplement: NAD3
- Active2 (Experimental): 812 mg dose of active
  Interventions: Dietary Supplement: NAD3
- Placebo (Placebo Comparator): placebo
  Interventions: Dietary Supplement: NAD3

INTERVENTIONS:
Dietary Supplement: NAD3 — NAD3 is an over-the-counter dietary supplement available online to consumers.

SUMMARY:
This is a randomized, parallel-group, placebo-controlled, clinical trial in middle-aged and older male and female subjects from Ohio. Subjects will take an over-the-counter dietary supplement or a placebo for 12 weeks. Outcome measures will include body weight, systolic and diastolic blood pressure, standard blood chemistries (e.g. chemistry panel, lipid panel, CBC with differential), changes in mood, vitality, energy, fatigue, productivity, digestive wellness (via anchored Visual Analogue Scales).

ELIGIBILITY:
Inclusion Criteria:

* Provide voluntary signed and dated informed consent.
* Be in good health as determined by medical history, physical, and routine blood chemistries.
* Age between the ages of 40 and 60 (inclusive).
* Body Mass Index (BMI) of 18.5-34.9 kg/m2 (normal to Class I obesity).
* Normotensive (supine, resting systolic blood pressure <140 mm Hg and diastolic blood pressure < 90 mm Hg. If the first measurement is slightly elevated above these limits, the subject will be given a brief (5 minute) rest period, and two more measurements will be taken. The average of all three measurements will be used to determine eligibility.
* Normal supine, resting heart rate (<90 per minute).
* Willing to duplicate their previous 24-hour diet, and fast for 10 hours prior each of the treatments.

Exclusion Criteria:

* History of uncontrolled diabetes.
* Regular use/consumption (i.e. at least 5 days/week) of resveratrol, quercetin, pterostilbene coQ10, grapefruit, nicotinamide riboside, probiotics, prebiotic fiber, green tea, niacin (vitamin B3), multivitamin/multimineral or products meant to promote "healthy aging" or "anti-aging" or "longevity" products in the 2 weeks prior to screening as well as throughout the study.
* Clinically significant abnormal blood work at screening.
* Consumption of > 2 alcoholic drinks per day.
* History of malignancy in the previous 5 years except for non-melanoma skin cancer (basal cell cancer or squamous cell cancer of the skin).
* Other known gastrointestinal or metabolic diseases that might impact nutrient absorption or metabolism, e.g. short bowel syndrome, diarrheal illnesses, history of colon resection, gastro paresis, Inborn-Errors-of-Metabolism (such as PKU).
* Chronic inflammatory condition/disease or unstable medical condition (e.g. rheumatoid arthritis, Crohn's disease, ulcerative colitis, Lupus, hepatitis, HIV/AIDS, etc.).
* Known sensitivity to any ingredient in the test formulations as listed in the Certificates-of-Analysis.
* Currently participating in another research study with an investigational product or have been in another research study in the past 30 days.
* History of drug or alcohol addiction or abuse within 1 year prior to screening.
* Treatment with any known enzyme-altering drugs such as barbiturates, glucocorticoids, macrolides, antidepressants, neuroleptics, imidazoles, or fluoroquinolones within 30 days prior to screening.
* Subjects who (for whatever reason) have been on a self-restricted diet, controlled diet or special therapeutic diet, or who have had substantial changes in eating habits within 30 days prior to screening.
* Donation of blood within 30 days or plasma within 7 days, prior to screening.
* History or presence of clinically significant diseases or conditions (e.g., cardiovascular, pulmonary, respiratory, hepatic, renal, hematological, gastrointestinal, endocrine, immunologic, dermatologic, neurological, or psychiatric) which, in the opinion of the medical staff, could confound the primary endpoints or place the subject at increased risk of harm if they were to participate.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2020-06-08 (Actual); Primary Completion 2021-01-29 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
body weight | baseline
  body weight in pounds
body weight | week 4
  body weight in pounds
body weight | week 8
  body weight in pounds
body weight | week 12
  body weight in pounds
blood pressure | baseline
  systolic and diastolic blood pressure in mm Hg
blood pressure | week 4
  systolic and diastolic blood pressure in mm Hg
blood pressure | week 8
  systolic and diastolic blood pressure in mm Hg
blood pressure | week 12
  systolic and diastolic blood pressure in mm Hg
blood lipids | baseline
  Cholesterol profile (concentration of total cholesterol, HDL, LDL, TAG)
blood lipids | week 4
  Cholesterol profile (concentration of total cholesterol, HDL, LDL, TAG)
blood lipids | week 8
  Cholesterol profile (concentration of total cholesterol, HDL, LDL, TAG)
blood lipids | week 12
  Cholesterol profile (concentration of total cholesterol, HDL, LDL, TAG)

SECONDARY OUTCOMES:
mood | baseline
  subjective measurement of mood (number rating from Likert style scale questionnaire)
mood | week 4
  subjective measurement of mood (number rating from Likert style scale questionnaire)
mood | week 8
  subjective measurement of mood (number rating from Likert style scale questionnaire)
mood | week 12
  subjective measurement of mood (number rating from Likert style scale questionnaire)
vitality | baseline
  subjective measurement of vitality (number rating from Likert style scale questionnaire)
vitality | week 4
  subjective measurement of vitality (number rating from Likert style scale questionnaire)
vitality | week 8
  subjective measurement of vitality (number rating from Likert style scale questionnaire)
vitality | week 12
  subjective measurement of vitality (number rating from Likert style scale questionnaire)
energy | baseline
  subjective measurement of energy (number rating from Likert style scale questionnaire)
energy | week 4
  subjective measurement of energy (number rating from Likert style scale questionnaire)
energy | week 8
  subjective measurement of energy (number rating from Likert style scale questionnaire)
energy | week 12
  subjective measurement of energy (number rating from Likert style scale questionnaire)

CONTACTS AND LOCATIONS:
Locations (1):
- The Center for Applied Health Sciences, Canfield, Ohio, United States